CLINICAL TRIAL: NCT05671432
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of CM326 Injection in the Treatment of Adult Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: The Study of CM326 in Moderate-to-severe Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM326-101102
Record Dates: First submitted 2022-12-26; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A: CM326, subcutaneous (SC)
  Interventions: Biological: CM326
- Group B (Experimental): Group A: CM326, subcutaneous (SC)
  Interventions: Biological: CM326
- Group C (Placebo Comparator): Group C: placebo, subcutaneous (SC)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CM326 — CM326 injection
  Arms: Group A; Group B
Other: Placebo — Placebo
  Arms: Group C

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled study to evaluate the efficacy, safety, tolerance, pharmacokinetics, pharmacodynamics, and immunogenicity of CM326 in moderate-severe atopic dermatitis subjects.

DETAILED DESCRIPTION:
The study consists of 3 periods, a up-to-4-week Screening Period, a 52-week Treatment Period and a 8-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* With confirmed Atopic Dermatitis (AD) at the screening.
* Age ≥ 18 years and ≤ 75 years, male or female.
* Have the ability to understand the nature of the study and voluntarily sign the informed consent.
* Be able to communicate well with investigators and follow up protocol requirements.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Received allergen specific immunotherapy (desensitization) within 6 months prior to baseline.
* Major surgery is planned during the study period.
* Women who are pregnant or breastfeeding, or who plan to become pregnant during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-12-27 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Eczema Area and Severity Index (EASI)-75 (≥75 percent reduction in EASI scores from baseline) at visit 16 | at week 16
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Proportion of patients with Investigator's Global Assessment (IGA) score = 0-1 and reduction from baseline of ≥2 points at Visit 16 | at week 16
  IGA is a 5-point scale ranging from 0 (clear) to 4 (very severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No